CLINICAL TRIAL: NCT04846790
Title: The Effect of a Combined Nature-based and Virtual Mindfulness Intervention on Perceived Stress in Healthcare Workers That Care for Patients With COVID-19
Brief Title: The Effect of a Combined Nature-based and Virtual Mindfulness Intervention on Perceived Stress in Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Ann Berger, M.D., Chief of the Pain and Palliative Care Service, National Institutes of Health Clinical Center (CC)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CC-000192
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Stress, Psychological; Sleep Disturbance; Burnout, Caregiver; Posttraumatic Stress Disorder; Anxiety; Depression
Keywords: Resilience; Mindfulness; Meditation; Nature; Interventions; COVID-19; Pandemic; Healthcare workers
MeSH Terms: conditions — Stress, Psychological; Parasomnias; Caregiver Burden; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a Phase III, randomized controlled trial, whereby ninety healthcare workers will be randomized into one of three groups: Nature+Mindfulness (n=30), Nature only (n=30), and Control (n=30).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study team members and participants will be blind to group allocation with the exception of one research assistant who will not be involved in providing the intervention to the participants or data analysis. There is no outcome assessor, outcomes will be self-reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): The control group will complete the first three assessments similar to the two treatment groups but will not participate in the nature-based or virtual mindfulness interventions. At the end of their study participation (~week 3), they will be offered the opportunity to partake in the nature-based and virtual mindfulness interventions.
- Nature Only (Active Comparator): The nature-based intervention is three days long, is offered at various locations throughout the United States, and includes activities such as hiking, mountain-biking, and kayaking. The healthcare workers can participate in the programs that are offered locally pending availability. Each program will enroll between 15 and 30 healthcare workers. All First Descents nature-based interventions have been intentionally designed with input from more than 450 hospital partners nationwide to improve psychosocial health, nurture supportive peer relationships, and better position healthcare workers to carry out their critical mission. There is no cost to attend, and meals and lodging are included. Special precautions against SARS-CoV-2 transmission are implemented.
  Interventions: Behavioral: Nature Only
- Nature+Mindfulness (Experimental): In the combined nature-based and virtual mindfulness intervention, participants will complete the nature intervention followed by the mindfulness intervention. The virtual mindfulness intervention is 10 days long and offered online. Each day the participant will receive a notification that a new mindfulness audio is ready for viewing, which is from 10 to 25 minutes long. Mindfulness exercises include mindful breathing, body scan, and loving-kindness meditation. Participants can view the daily audio as many times as they wish but cannot view the next day's content to maintain treatment fidelity. At the end of each day, participants will be asked to indicate if they viewed the mindfulness audio to track adherence.
  Interventions: Behavioral: Nature+Mindfulness

INTERVENTIONS:
Behavioral: Nature Only — See above for description.
  Arms: Nature Only
Behavioral: Nature+Mindfulness — See above for description.
  Arms: Nature+Mindfulness

SUMMARY:
Rationale: Healthcare workers that care for patients with COVID-19 are at increased risk for stress-related symptoms. When these symptoms are chronic, they can result in burnout and other mental health conditions that can exacerbate the current national health crisis. Social distancing can limit the accessibility of mental health services. Feasible and effective interventions are needed to reduce stress-related symptoms and promote resilience in this population, while adhering to federal and local guidelines to mitigate the transmission of SARS-CoV-2.

Objectives: To investigate the feasibility and efficacy of a combined nature-based and virtual mindfulness intervention on stress-related symptoms and psychological resilience in healthcare workers that care for patients with COVID-19. Both components are reported to reduce levels of perceived stress and increase psychological resilience; however, the potential additive effect of their combined delivery is unknown.

Methods: Ninety healthcare workers will be randomized into one of three groups: Nature+Mindfulness (n=30), Nature only (n=30), and Control (n=30). All participants will undergo assessments at baseline (week 0), post nature intervention (~week 1), and post mindfulness intervention (~week 3). The two intervention groups will have one final assessment at 2-month follow-up (~week 11). Perceived stress is the primary endpoint and will be assessed with the Perceived Stress Scale. Secondary endpoints include sleep quality, burnout, posttraumatic stress, anxiety, depression, mindfulness, self-efficacy, and psycho-social-spiritual healing.

Anticipated Results: We anticipate that participants in the Nature+Mindfulness group will have greater reductions in stress-related symptoms and greater increases in psychological resilience compared with the Nature only and Control groups.

DETAILED DESCRIPTION:
Potential participants will be recruited through First Descents, a non-profit 501(c)(3) organization located in the United States.

The nature-based intervention is three days long and includes activities such as hiking, mountain-biking, and kayaking. The virtual mindfulness intervention is 10 to 25 minutes daily for 10 days and is offered online. Mindfulness exercises include mindful breathing, body scan, and loving-kindness meditation.

ELIGIBILITY:
Inclusion: In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Is 18 years old or older
2. Is a healthcare worker that cares for patients with COVID-19
3. Has access to technology to access study resources online
4. Is fluent in English
5. Is able to provide their own consent

Exclusion: An individual who meets any of the following criteria will be excluded from participation in this study:

1. Is experiencing an acute psychiatric condition
2. Has a hearing impairment that is not modified with aids or devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline (week 0), Post Nature Intervention (week 1), Post Mindfulness Intervention (week 3), Follow-up (week 11)
  The Perceived Stress Scale (PSS) is used to assess self-reported perceived stress. It is a 10-item scale, with a total range from 0 (no symptoms) to 40 (highest severity).

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline (week 0), Post Nature Intervention (week 1), Post Mindfulness Intervention (week 3), Follow-up (week 11)
  The Insomnia Severity Index (ISI) is used to assess self-reported sleep quality. It is a 7-item index, with a total range from 0 (no symptoms) to 28 (highest severity).
Maslach Burnout Inventory (MBI 2-Item) | Baseline (week 0), Post Nature Intervention (week 1), Post Mindfulness Intervention (week 3), Follow-up (week 11)
  The Maslach Burnout Inventory (MBI 2-Item) is used to assess self-reported burnout. The 2-Item inventory assesses emotional exhaustion and depersonalization separately from 1 (no symptoms) to 7 (highest severity).
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline (week 0), Post Nature Intervention (week 1), Post Mindfulness Intervention (week 3), Follow-up (week 11)
  The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) is used to assess self-reported posttraumatic stress symptoms. It is a 20-item checklist, with a total range from 20 (no symptoms) to 100 (highest severity).
Hospital Anxiety and Depression Scale (HADS) | Baseline (week 0), Post Nature Intervention (week 1), Post Mindfulness Intervention (week 3), Follow-up (week 11)
  The Hospital Anxiety and Depression Scale (HADS) is used to assess self-reported anxiety and depression. It consists of two 7-item scales (for anxiety and for depression), with a sub-scale range from 0 (no symptoms) to 21 (highest severity).
Mindful Attention Awareness Scale-State Version (MAAS-S) | Baseline (week 0), Post Nature Intervention (week 1), Post Mindfulness Intervention (week 3), Follow-up (week 11)
  The Mindful Attention Awareness Scale-State Version (MAAS-S) is used to assess self-reported state mindfulness. It is a 5-item scale, with a total range from 0 (high mindfulness) to 30 (low mindfulness).
General Self-Efficacy Scale (GSF) | Baseline (week 0), Post Nature Intervention (week 1), Post Mindfulness Intervention (week 3), Follow-up (week 11)
  The General Self-Efficacy Scale (GSF) is used to assess self-reported coping ability in daily life. It is a 10-item scale, with a total range from 10 (low self-efficacy) to 40 (high self-efficacy).
National Institutes of Health-Healing Experience of All Life Stressors (NIH-HEALS) | Baseline (week 0), Post Nature Intervention (week 1), Post Mindfulness Intervention (week 3), Follow-up (week 11)
  The National Institutes of Health-Healing Experience of All Life Stressors (NIH-HEALS) is used to assess self-reported psycho-social-spiritual mechanisms for coping. It is a 35-item questionnaire, with a total range from 35 (low coping) to 175 (high coping).

CONTACTS AND LOCATIONS:
Overall Officials: Ann Berger, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institutes of Health, Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ameli R, Sinaii N, West CP, Luna MJ, Panahi S, Zoosman M, Rusch HL, Berger A. Effect of a Brief Mindfulness-Based Program on Stress in Health Care Professionals at a US Biomedical Research Hospital: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2013424. doi: 10.1001/jamanetworkopen.2020.13424. PMID 32840621
- [Background] Rusch HL, Rosario M, Levison LM, Olivera A, Livingston WS, Wu T, Gill JM. The effect of mindfulness meditation on sleep quality: a systematic review and meta-analysis of randomized controlled trials. Ann N Y Acad Sci. 2019 Jun;1445(1):5-16. doi: 10.1111/nyas.13996. Epub 2018 Dec 21. PMID 30575050
- [Background] Ameli R, Sinaii N, Luna MJ, Cheringal J, Gril B, Berger A. The National Institutes of Health measure of Healing Experience of All Life Stressors (NIH-HEALS): Factor analysis and validation. PLoS One. 2018 Dec 12;13(12):e0207820. doi: 10.1371/journal.pone.0207820. eCollection 2018. PMID 30540764
- [Background] Ameli R, Skeath P, Abraham PA, Panahi S, Kazman JB, Foote F, Deuster PA, Ahmad N, Berger A. A nature-based health intervention at a military healthcare center: a randomized, controlled, cross-over study. PeerJ. 2021 Jan 4;9:e10519. doi: 10.7717/peerj.10519. eCollection 2021. PMID 33505785